CLINICAL TRIAL: NCT05166811
Title: Intravenous Magnesium: Prompt Use for Asthma in Children Treated in the Emergency Department
Brief Title: Timely Intravenous Magnesium for Asthma in Children
Acronym: IMPACT-ED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Nationwide Children's Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mike Johnson, Associate Professor of Pediatrics, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 104082; 1R34HL152047-01A1 (NIH)
Record Dates: First submitted 2021-11-23; First posted 2021-12-22 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Asthma
Keywords: asthma; IV Magnesium
MeSH Terms: conditions — Asthma | interventions — Magnesium Sulfate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Doses will be prepared ahead of time by an investigational pharmacist, arms will be identical in appearance, and clinicians administering the study drug will be blinded to the study arm the patient receives.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 75 mg/kg (Active Comparator): Doses for each IVMg arm will be prepared in identical manner, by drawing a specified volume of IVMg from the commercial container using sterile technique and mixing in a polyvinylchloride container with a specified volume of sterile water. For the 75 mg/kg arm, this will be accomplished by mixing 37.5 mL of IVMg (80 mg/mL) with 2.5 mL of sterile water for a final concentration of 75 mg/mL and volume of 40 mL. After randomization the institutional pharmacist will draw dosages (1 mL/kg, with max of 40 mL) from previously prepared vials. The dose will be delivered by the clinical nurse over 20 minutes through a peripheral IV.
  Interventions: Drug: Magnesium Sulfate, Heptahydrate
- 50 mg/kg (Active Comparator): Doses for each IVMg arm will be prepared in identical manner, by drawing a specified volume of IVMg from the commercial container using sterile technique and mixing in a polyvinylchloride container with a specified volume of sterile water. For the 50 mg/kg arm, this will be accomplished by mixing 25 mL of IVMg (80 mg/mL) with 15 mL of sterile water for a final concentration of 50 mg/mL and volume of 40 mL. After randomization the institutional pharmacist will draw dosages (1 mL/kg, with max of 40 mL) from previously prepared vials. The dose will be delivered by the clinical nurse over 20 minutes through a peripheral IV.
  Interventions: Drug: Magnesium Sulfate, Heptahydrate
- Placebo (Placebo Comparator): For the placebo arm, 40 mL of 0.9% sodium chloride solution will be drawn into a polyvinylchloride container identical in appearance to the containers used for the IVMg arms. After randomization the institutional pharmacist will draw dosages (1 mL/kg, with max of 40 mL) from previously prepared vials. The dose will be delivered by the clinical nurse over 20 minutes through a peripheral IV.
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Magnesium Sulfate, Heptahydrate — A single dose of intravenous magnesium sulfate given over 20 minutes through a peripheral intravenous line. Two arms of the study will deliver intravenous magnesium, one at a dose of 50 mg/kg, and the other at a dose of 75 mg/kg.
  Other Names: Intravenous magnesium sulfate
  Arms: 50 mg/kg; 75 mg/kg
Drug: 0.9% saline — A single dose of intravenous 0.9% sodium chloride given over 20 minutes through a peripheral intravenous line as the placebo arm of the study.
  Other Names: normal saline; 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
Many children currently being hospitalized with severe asthma could potentially avoid hospitalization and be sent home if their treatment in the emergency department was more effective. The investigators will conduct a pilot trial that will lead to a larger study to conclusively answer whether a simple and inexpensive medicine, intravenous magnesium sulfate, can be used in the emergency department to prevent hospitalization for these children.

DETAILED DESCRIPTION:
5.4.1 Acquisition The specific study agent to be used in this pilot trial is Magnesium Sulfate in Water for Injection, a sterile, nonpyrogenic solution of magnesium sulfate heptahydrate in water. Study agent will be acquired by each hospital's research pharmacy from Pfizer, Inc as a solution of magnesium sulfate in water at 80 mg/mL. Agent will be shipped directly from Pfizer to each study hospital pharmacy.

5.4.2 Preparation, Storage & Labeling Doses for each IVMg arm will be prepared in identical manner, by drawing a specified volume of Intravenous Magnesium Sulfate (IVMg) from the commercial container using sterile technique and mixing in a polyvinylchloride container with a specified volume of sterile water. For the 50 mg/kg arm, this will be accomplished by mixing 25 mL of IVMg (80 mg/mL) with 15 mL of sterile water for a final concentration of 50 mg/mL and volume of 40 mL. For the 75 mg/kg arm, this will be accomplished by mixing 37.5 mL of IVMg (80 mg/mL) with 2.5 mL of sterile water for a final concentration of 75 mg/mL and volume of 40 mL. For the placebo arm, 40 mL of 0.9% sodium chloride solution will be drawn into a polyvinylchloride container identical in appearance to the containers used for the IVMg arms. Each prepared dose will be labeled according to the sequential randomization scheme and stored according to local pharmacy procedure. Unused doses prepared locally will be replaced after one week of storage.

5.4.3 Dosing Schedule

After randomization the institutional pharmacist will draw equivolumetric dosages (1 mL/kg, with max of 40 mL) from previously prepared vials. Enrolled subjects will be randomized to one of three arms:

* IVMg 75 mg/kg arm: 75 mg/kg (max 3 gm) infused over 20 minutes through a peripheral IV catheter
* IVMg 50 mg/kg arm: 50 mg/kg (max 2 gm) infused over 20 minutes through a peripheral IV catheter
* Placebo arm: 1 mL/kg (max 40 ml) of normal saline over 20 minutes through a peripheral IV catheter 5.4.4 Dose Modification for Potential Toxicity Clinicians will not administer IVMg to enrolled subjects outside of the study protocol until study outcomes have been determined 2 hours after the start of the infusion. The half-life of IVMg is approximately 2 hours.49 Repeated-dose protocols in an ICU setting that gave as much as 125 mg/kg IVMg to children with asthma over two hours produced no hypotension or other serious adverse effects.47 Because of this margin of safety, open-label IVMg 50 mg/kg can be administered safely 2 hours after the study infusion under strict study monitoring protocols without need for unblinding.

ELIGIBILITY:
Inclusion criteria are:

1. A prior physician diagnosis of asthma confirmed by a treating physician in the ED who has spoken with the patient and family and reviewed the medical record (ED attending or fellow physician)
2. Severe acute asthma, defined as a Pediatric Respiratory Assessment Measure (PRAM) score of 7 or greater as assessed by a treating physician at the time of screening using the study scoring instrument, which takes 60 seconds to complete
3. Children 2-17 years of age

Exclusion criteria are:

* Known pregnancy (by patient or parent report) or positive pregnancy test on females 12 years of age and older
* Age-adjusted hypotension at presentation using age-based Pediatric Advanced Life Support parameters (children >1 year to 10 years, systolic blood pressure (SBP)<(70 + 2 x age in years); >10 years, SBP < 90 mmHg)71
* Known severe renal impairment (by parent or patient report)
* Application of assisted ventilation before enrollment assessment (intubated, bi-level positive airway pressure, continuous positive airway pressure)
* Received IVMg within 24 hours prior to screening (by parent or patient report or medical record review)
* Enrollment assessment is 60 minutes after the start of ED treatment (start of first albuterol treatment)
* Previous enrollment in the same trial (by research coordinator review of trial records)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Primary Children's Hospital, Salt Lake City, Utah

REFERENCES:
- [Derived] Johnson MD, Barney BJ, Rower JE, Finkelstein Y, Zorc JJ. Intravenous Magnesium: Prompt Use for Asthma in Children Treated in the Emergency Department (IMPACT-ED): Protocol for a Multicenter Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Jul 17;12:e48302. doi: 10.2196/48302. PMID 37459153

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at three sites within the Pediatric Emergency Care Applied Research Network (PECARN). The three enrolling sites are EDs at tertiary pediatric hospitals and are geographically and demographically diverse. Eligible participants were identified from children presenting to the ED for treatment of acute asthma. Screening occurred at sites from September 2022 through May 2023.
Groups:
- 50 mg/kg: Doses for each intravenous magnesium sulfate (IVMg) arm will be prepared in identical manner, by drawing a specified volume of IVMg from the commercial container using sterile technique and mixing in a polyvinylchloride container with a specified volume of sterile water. For the 50 mg/kg arm, this will be accomplished by mixing 25 mL of IVMg (80 mg/mL) with 15 mL of sterile water for a final concentration of 50 mg/mL and volume of 40 mL. After randomization the institutional pharmacist will draw dosages (1 mL/kg, with max of 40 mL) from previously prepared vials. The dose will be delivered by the clinical nurse over 20 minutes through a peripheral IV.
  Magnesium Sulfate, Heptahydrate: A single dose of intravenous magnesium sulfate given over 20 minutes through a peripheral intravenous line.
- 75 mg/kg: Doses for each intravenous magnesium sulfate (IVMg) arm will be prepared in identical manner, by drawing a specified volume of IVMg from the commercial container using sterile technique and mixing in a polyvinylchloride container with a specified volume of sterile water. For the 75 mg/kg arm, this will be accomplished by mixing 37.5 mL of IVMg (80 mg/mL) with 2.5 mL of sterile water for a final concentration of 75 mg/mL and volume of 40 mL. After randomization the institutional pharmacist will draw dosages (1 mL/kg, with max of 40 mL) from previously prepared vials. The dose will be delivered by the clinical nurse over 20 minutes through a peripheral IV.
  Magnesium Sulfate, Heptahydrate: A single dose of intravenous magnesium sulfate given over 20 minutes through a peripheral intravenous line.
Period: Overall Study
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Started (Participants enrolled in study) | 18 | 17 | 17
Completed (Participants randomized to study arm) | 18 | 17 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: For the placebo arm, 40 mL of 0.9% sodium chloride solution was drawn into a polyvinylchloride container identical in appearance to the containers used for the IVMg arms. After randomization the institutional pharmacist prepared the dosage (1 mL/kg, with max of 40 mL) from previously prepared container. The dose was delivered by the clinical nurse over 20 minutes through a peripheral IV.
  0.9% saline: A single dose of intravenous 0.9% sodium chloride given over 20 minutes through a peripheral intravenous line as the placebo arm of the study.
- 50 mg/kg: Doses for each IVMg arm were prepared in identical manner, by drawing a specified volume of IVMg from the commercial container using sterile technique and mixing in a polyvinylchloride container with a specified volume of sterile water. For the 50 mg/kg arm, this was accomplished by mixing 25 mL of IVMg (80 mg/mL) with 15 mL of sterile water for a final concentration of 50 mg/mL and volume of 40 mL. After randomization the institutional pharmacist prepared the dosage (1 mL/kg, with max of 40 mL) from previously prepared container. The dose was delivered by the clinical nurse over 20 minutes through a peripheral IV.
  Magnesium Sulfate, Heptahydrate: A single dose of intravenous magnesium sulfate given over 20 minutes through a peripheral intravenous line.
- 75 mg/kg: Doses for each IVMg arm were prepared in identical manner, by drawing a specified volume of IVMg from the commercial container using sterile technique and mixing in a polyvinylchloride container with a specified volume of sterile water. For the 75 mg/kg arm, this was accomplished by mixing 37.5 mL of IVMg (80 mg/mL) with 2.5 mL of sterile water for a final concentration of 75 mg/mL and volume of 40 mL. After randomization the institutional pharmacist prepared the dosage (1 mL/kg, with max of 40 mL) from previously prepared container. The dose was by the clinical nurse over 20 minutes through a peripheral IV.
  Magnesium Sulfate, Heptahydrate: A single dose of intravenous magnesium sulfate given over 20 minutes through a peripheral intravenous line.
- Total: Total of all reporting groups
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg | Total
Number analyzed (Participants) | 18 | 17 | 17 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.0 (5.9) | 7.4 (7.4) | 7.3 (4.3) | 7.3 (6.4)
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 5.9 [4.6 to 9.3] | 7.4 [5.3 to 9.9] | 5.8 [3.9 to 11.2] | 6.4 [4.2 to 9.7]
Age, Customized [Count of Participants; unit: Participants]
  Age Group: 2-4 years | 7 | 4 | 6 | 17
  Age Group: 5-17 years | 10 | 12 | 11 | 33
  Age Group: Unknown | 1 | 1 | 0 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 12 | 11 | 12 | 35
  Sex: Female | 5 | 5 | 5 | 15
  Sex: Unknown | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 0 | 8
  Not Hispanic or Latino | 13 | 11 | 16 | 40
  Unknown or Not Reported | 2 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 5 | 8 | 6 | 19
  White | 10 | 6 | 4 | 20
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 1 | 2 | 2 | 5
Weight [Mean (Standard Deviation); unit: kilograms] | 28 (16.4) | 32.7 (21.3) | 27.7 (19.7) | 29.4 (18.9)
Prior hospitalizations for asthma [Count of Participants; unit: Participants] | 9 | 12 | 14 | 35
ED visit for asthma in the last 12 months [Count of Participants; unit: Participants] | 9 | 12 | 14 | 35
Prescribed a daily controller medication [Count of Participants; unit: Participants] | 18 | 17 | 17 | 52
Taking controller medication 4+ days a week [Count of Participants; unit: Participants] | 8 | 10 | 7 | 25
Personal history of eczema [Count of Participants; unit: Participants] | 8 | 9 | 6 | 23
Personal history of anaphylaxis [Count of Participants; unit: Participants] | 2 | 2 | 1 | 5
Personal history of prematurity [Count of Participants; unit: Participants] | 5 | 2 | 5 | 12
Parent with asthma [Count of Participants; unit: Participants] | 12 | 10 | 12 | 34
Parent with eczema [Count of Participants; unit: Participants] | 6 | 8 | 8 | 22
Parent with seasonal allergies [Count of Participants; unit: Participants] | 10 | 11 | 12 | 33
Arrival pulse oximeter reading 95% or higher [Count of Participants; unit: Participants] | 4 | 5 | 4 | 13
Arrival pulse oximeter reading 92-94% [Count of Participants; unit: Participants] | 5 | 5 | 6 | 16
Arrival pulse oximeter reading 91% or lower [Count of Participants; unit: Participants] | 9 | 7 | 7 | 23
Weight [Median (Inter-Quartile Range); unit: kilograms] | 20.8 [17.0 to 35.9] | 28.4 [19.6 to 34.1] | 18.1 [16.5 to 31.7] | 21.1 [17.1 to 34.9]

OUTCOME MEASURES:

1. Primary Outcome: Enrollment
Description: The primary outcome in this pilot trial is demonstration of the ability to enroll severely ill children with asthma in a randomized trial requiring timely delivery of IVMg or placebo. The investigators anticipate that the primary outcome of the future large trial will be the proportion of children hospitalized at the index visit in each arm.
Time Frame: 7 months of enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 17 | 17
Participants | 18 | 17 | 17

2. Secondary Outcome: Hospitalization
Description: Actual patient disposition from medical record review after completion of ED treatment. Hospitalization will be defined as any outcome other than discharge from the ED, including hospitalization in an ICU, hospital unit, or observation area.
Time Frame: Actual disposition from chart review 1 week after enrollment.
Population: Participants who were enrolled were included in the intention-to-treat (ITT) population regardless of whether they received study drug according to their randomization arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 17 | 17
Participants | 12 | 12 | 14

3. Secondary Outcome: Hospitalization Anticipated by Treating Physician 2 Hours After Start of Study Infusion
Description: The treating clinician's stated disposition two hours after the start of study infusion.
Time Frame: Physician-anticipated hospitalization 2 hours after the start of study drug infusion
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 17 | 17
Participants | 13 | 12 | 13

4. Secondary Outcome: Adverse Events and Safety Profiles - Hypotension and Perfusion
Description: Decrease in blood pressure was categorized based on degree of associated symptoms and defined as occurring less than 2 hours after the start of study drug infusion or 2 hours and later. Hypotension is defined by age-based Pediatric Advanced Life Support guidelines.
Time Frame: 2 hours after study drug infusion.
Population: Participants in whom the study drug infusion was started were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
Participants
  Hypotension within 2 hours of start of study infusion | 2 | 1 | 1
  Hypotension more than 2 hours after start of study infusion | 2 | 4 | 3
  Poor perfusion during hypotension within 2 hours of start of study infusion | 0 | 0 | 0
  No hypotension measured | 14 | 11 | 11

5. Secondary Outcome: Rescue Therapies Used During ED Care - SQ or IM Epinephrine
Description: Count of the number of participants that were administered subcutaneous (SQ) or intramuscular (IM) epinephrine while in the ED during the index visit, recorded by chart review approximately one week after enrollment.
Time Frame: One week after enrollment
Population: Participants who were enrolled were included in the intention-to-treat (ITT) population for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 17 | 17
Participants
  SQ or IM epinephrine | 1 | 1 | 0
  not administered SQ or IM epinephrine | 17 | 16 | 17

6. Secondary Outcome: Return ED Visit
Description: In patients discharged from the ED, any ED visit and/or hospitalization following discharge.
Time Frame: Within 10 days after ED discharge
Population: Participants who were enrolled were included in the intention-to-treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 17 | 17
Participants | 5 | 0 | 1

7. Secondary Outcome: Baseline Serum Magnesium
Time Frame: At IV placement before infusion of study drug
Population: Participants in whom the study drug infusion was started were included in the safety population used for these results.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
mg/dL | 1.95 (0.13) | 1.95 (0.23) | 2.20 (0.55)

8. Secondary Outcome: Baseline Ionized Magnesium
Time Frame: At IV placement before infusion of study drug
Population: Participants in whom the study drug infusion was started were included in the safety population used for these results.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
mg/dL | 0.57 (0.04) | 0.57 (0.10) | 0.70 (0.24)

9. Secondary Outcome: Post-infusion Serum Magnesium 1
Time Frame: 20-40 minutes after the start of study drug infusion
Population: Participants in whom the study drug infusion was started were included in the safety population used for these results.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 16 | 16 | 15
mg/dL | 1.86 (0.20) | 4.13 (3.32) | 3.79 (0.92)

10. Secondary Outcome: Post-infusion Ionized Magnesium 1
Time Frame: 20-40 minutes after the start of study drug infusion
Population: Participants in whom the study drug infusion was started were included in the safety population used for these results.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 16 | 16 | 15
mg/dL | 0.54 (0.05) | 1.06 (0.25) | 1.15 (0.24)

11. Secondary Outcome: Post-infusion Serum Magnesium 2
Time Frame: 90-150 minutes after the start of study drug infusion
Population: Participants in whom the study drug infusion was started were included in the safety population used for these results.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 14 | 14 | 14
mg/dL | 1.91 (0.14) | 2.54 (0.24) | 2.84 (0.21)

12. Secondary Outcome: Post-infusion Ionized Magnesium 2
Time Frame: 90-150 minutes after the start of study drug infusion
Population: Participants in whom the study drug infusion was started were included in the safety population used for these results.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 14 | 14 | 14
mg/dL | 0.57 (0.04) | 0.76 (0.09) | 0.85 (0.12)

13. Secondary Outcome: Rescue Therapies Used During ED Care - IV Epinephrine
Description: Count of the number of participants that were administered intravenous (IV) epinephrine while in the ED during the index visit, recorded by chart review approximately one week after enrollment.
Time Frame: One week after enrollment
Population: Participants who were enrolled were included in the intention-to-treat (ITT) population for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 17 | 17
Participants
  IV epinephrine | 0 | 0 | 0
  not administered IV epinephrine | 18 | 17 | 17

14. Secondary Outcome: Rescue Therapies Used During ED Care - IV Terbutaline
Description: Count of the number of participants that were administered intravenous (IV) terbutaline while in the ED during the index visit, recorded by chart review approximately one week after enrollment.
Time Frame: One week after enrollment
Population: Participants who were enrolled were included in the intention-to-treat (ITT) population for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 17 | 17
Participants
  IV terbutaline | 0 | 0 | 0
  not administered IV terbutaline | 18 | 17 | 17

15. Secondary Outcome: Rescue Therapies Used During ED Care - IV Magnesium
Description: Count of the number of participants that were administered intravenous (IV) magnesium while in the ED during the index visit aside from any study infusion administered, recorded by chart review approximately one week after enrollment.
Time Frame: One week after enrollment
Population: Participants who were enrolled were included in the intention-to-treat (ITT) population for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 17 | 17
Participants
  IV magnesium | 2 | 2 | 4
  not administered IV magnesium | 16 | 15 | 13

16. Secondary Outcome: Adverse Events and Safety Profiles - Supraventricular Tachycardia
Description: Adverse events were assessed through chart review and phone call with the parent of the participant one week after enrollment. Timing after start of study infusion was not recorded.
Time Frame: 1 week
Population: Participants in whom the study drug infusion was started were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
Participants
  supraventricular tachycardia | 0 | 0 | 1
  No supraventricular tachycardia | 18 | 16 | 14

17. Secondary Outcome: Adverse Events and Safety Profiles - Abdominal Discomfort
Description: as for outcome 16
Time Frame: 1 week
Population: Participants in whom the study drug infusion was started were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
Participants
  abdominal discomfort | 0 | 0 | 1
  no abdominal discomfort | 18 | 16 | 14

18. Secondary Outcome: Adverse Events and Safety Profiles - Vomiting
Description: as for outcome 16
Time Frame: 1 week
Population: Participants in whom the study drug infusion was started were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
Participants
  vomiting | 0 | 0 | 1
  no vomiting | 18 | 16 | 14

19. Secondary Outcome: Adverse Events and Safety Profiles - Fatigue
Description: as for outcome 16
Time Frame: 1 week
Population: Participants in whom the study drug infusion was started were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
Participants
  fatigue | 0 | 1 | 0
  no fatigue | 18 | 15 | 15

20. Secondary Outcome: Adverse Events and Safety Profiles - Hypokalemia
Description: as for outcome 16
Time Frame: 1 week
Population: Participants in whom the study drug infusion was started were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
Participants
  hypokalemia | 0 | 1 | 0
  no hypokalemia | 18 | 15 | 15

21. Secondary Outcome: Adverse Events and Safety Profiles - Delirium
Description: as for outcome 16
Time Frame: 1 week
Population: Participants in whom the study drug infusion was started were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
Participants
  delirium | 0 | 0 | 1
  no delirium | 18 | 16 | 14

22. Secondary Outcome: Adverse Events and Safety Profiles - Hypoxia
Description: as for outcome 16
Time Frame: 1 week
Population: Participants in whom the study drug infusion was started were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
Participants
  hypoxia | 1 | 1 | 2
  no hypoxia | 17 | 15 | 13

23. Secondary Outcome: Adverse Events and Safety Profiles - Respiratory Distress
Description: as for outcome 16
Time Frame: 1 week
Population: Participants in whom the study drug infusion was started were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
Participants
  respiratory distress | 2 | 0 | 0
  no respiratory distress | 16 | 16 | 15

24. Secondary Outcome: Adverse Events and Safety Profiles - Metabolic Acidosis
Description: as for outcome 16
Time Frame: 1 week
Population: Participants in whom the study drug infusion was started were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
Participants
  metabolic acidosis | 1 | 0 | 0
  no metabolic acidosis | 17 | 16 | 15

25. Secondary Outcome: Adverse Events and Safety Profiles - Duodenal Ulcer Perforation
Description: as for outcome 16
Time Frame: 1 week
Population: Participants in whom the study drug infusion was started were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
Number analyzed (Participants) | 18 | 16 | 15
Participants
  duodenal ulcer perforation | 1 | 0 | 0
  no duodenal ulcer perforation | 17 | 16 | 15

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated 1 week after enrollment through review of the medical record and phone call with parent of the participant.
Description: No different that expected definitions.
Arm/Group | Placebo | 50 mg/kg | 75 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/18 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 4/18 | 5/16 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | 50 mg/kg (N=16) | 75 mg/kg (N=15)
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — During treatment in the Emergency Department, the patient had persistent severe symptoms. The patient had some improvement of respiratory distress on BiPAP and was transferred to the pediatric ICU.
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — The patient had worsening respiratory distress after hospitalization, and was given additional doses of IV mag and was placed on continuous albuterol.
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | 50 mg/kg (N=16) | 75 mg/kg (N=15)
supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
hypokalemia (General disorders) | 0 (0) | 1 (1) | 0 (0)
delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
hypotension (Cardiac disorders) | 2 (2) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT05166811/Prot_SAP_002.pdf
  • Informed Consent Form: Parental Permission (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT05166811/ICF_000.pdf
  • Informed Consent Form: Assent (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT05166811/ICF_001.pdf